CLINICAL TRIAL: NCT03082222
Title: An Open, Multicentric, Non-Interventional Observational Study Investigating Retention, Seizure Control and Tolerability in Epilepsy Patients With Partial Onset Seizures Receiving Eslicarbazepine Acetate (ESL) in Different Therapy Situations
Brief Title: ZEDEBAC: Zebinix Effects in Dependency of Baseline Conditions
Status: Completed | Type: Observational
Sponsor: Eisai GmbH (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: E2093-M044-405
Record Dates: First submitted 2017-02-21; First posted 2017-03-17 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-08

CONDITIONS: Focal Epilepsy
Keywords: partial onset seizures with or without secondary generalization
MeSH Terms: conditions — Epilepsies, Partial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Group 1: Participants with epilepsy, partial onset seizures with or without secondary generalization with one concomitant antiepileptic drug (AED) at baseline
- Group 2: Participants with epilepsy, partial onset seizures with or without secondary generalization with two or more concomitant AEDs at baseline
- Group 3: Participants with epilepsy, partial onset seizures with or without secondary generalization with eslicarbazepine acetate (ESL) as anticonvulsant monotherapy

SUMMARY:
This is a non interventional prospective study. Centers will enroll adult participants with partial onset seizures with or without secondary generalisation for whom the clinician has decided to initiate eslicarbazepine acetate (ESL) as an adjunctive therapy or monotherapy prior to the decision to take part in this study. Participants to be enrolled into the study will receive ESL either as an adjunctive therapy to one baseline antiepileptic drug (AED) or to at least two baseline AEDs or as monotherapy. Participants will be seen at baseline and at a follow-up visit after approximately 6 months to assess retention, efficacy, tolerability, quality of life (optional), and cognitive performances (optional).

ELIGIBILITY:
Inclusion Criteria:

1. Partial onset seizures with or without secondary generalisation in conjunction with a diagnosed epilepsy of symptomatic or unknown course.
2. The decision to prescribe Eslicarbazepine acetate (ESL) was taken independent of and prior to enrollment into this study.
3. Treatment with ESL is in agreement with the valid summary of product characteristics (SmPC) version, particularly with the licensed indication.
4. Age 18 years and older.
5. Participant's written consent.

Exclusion Criteria:

1. Known psychogenic non-epileptic attacks.
2. Participation in an interventional study.
3. Previous enrollment in the current study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible participants appearing to their treating physician or clinic for routine visits will be invited to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-10-29 (Actual); Study Completion 2018-10-29 (Actual)

PRIMARY OUTCOMES:
Percentage of participants continuing treatment with Eslicarbazepine Acetate (ESL) | At follow-up visit (occurring after approximately 6 months of treatment)

SECONDARY OUTCOMES:
Change from baseline in total seizure frequency | Baseline (the 3 months period prior to initiation of treatment with ESL) and 3 months period prior to follow-up visit (occurring after approximately 6 months of treatment)
Change from baseline in seizure frequency by seizure type | Baseline (the 3 months period prior to initiation of treatment with ESL) and 3 months period prior to follow-up visit (occurring after approximately 6 months of treatment)
Responder Rate | Baseline (the 3 months period prior to initiation of treatment with ESL) and 3 months period prior to follow-up visit (occurring after approximately 6 months of treatment)
  Percentage of participants achieving a reduction in total seizure frequency by at least 50% within the 3-month period prior to Follow-Up in comparison with Baseline (the 3-month period prior to initiation of treatment with ESL)
Percentage of participants achieving seizure free state | 3 months period prior to follow-up visit (occurring after approximately 6 months of treatment)
Change from baseline in Quality of Life in Epilepsy Inventory-10 (QOLIE-10) | Baseline (the 3 months period prior to initiation of treatment with ESL) and 3 months period prior to follow-up visit (occurring after approximately 6 months of treatment)
  Only in centers where this questionnaire is part of the clinical routine.
Change from baseline in NeuroCog FX subset scores | Baseline (the 3 months period prior to initiation of treatment with ESL) and at follow-up visit (occurring after approximately 6 months of treatment)
Percentage of participants with Adverse Events (AEs) | From signing of informed consent up to the follow-up visit (occurring after approximately 6 months of treatment)

CONTACTS AND LOCATIONS:
Locations (1):
- Multiple Locations, Germany